CLINICAL TRIAL: NCT03503734
Title: Integrated Care for Migraine and Chronic Tension-type Headaches
Acronym: IV
Status: Completed | Type: Observational
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, Research Director, Universität Duisburg-Essen
Other Study IDs: 11-4749
Record Dates: First submitted 2018-04-11; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Chronic Headache
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Integrated headache care: The treatment can be realized on an inpatient, outpatient and/or day care basis, according to the severity level of illness and comorbidities.
  The inpatient treatment takes place at the Department of Internal and Integrative Medicine. The stay is slated for 14 days.
  Day care can follow the inpatient stay or can be applied as sole therapy. As part of the standard care provided at the Department for Internal and Integrative Medicine, it occurs at a semi-residential clinic for 6 hours once a week over a total of 10 weeks.
  The outpatient treatment is delivered in the Department's outpatient ward. It consists of acupuncture, cupping, hydrotherapy and massages as well as nutritional counseling. The patients can additionally be offered one-to-one mind-body-medicine interventions.
  Interventions: Behavioral: Integrated headache care

INTERVENTIONS:
Behavioral: Integrated headache care — The treatment can be realized on an inpatient, outpatient and/or day care basis, according to the severity level of illness and comorbidities.
  The inpatient treatment takes place at the Department of Internal and Integrative Medicine. The stay is slated for 14 days.
  Day care can follow the inpatient stay or can be applied as sole therapy. As part of the standard care provided at the Department for Internal and Integrative Medicine, it occurs at a semi-residential clinic for 6 hours once a week over a total of 10 weeks.
  The outpatient treatment is delivered in the Department's outpatient ward. It consists of acupuncture, cupping, hydrotherapy and massages as well as nutritional counseling. The patients can additionally be offered one-to-one mind-body-medicine interventions.

SUMMARY:
Chronic headache is among the most common neurological disorders with major physical, psychological, social and economic impact. The aim of this prospective observational study isto investigate the effects of an interdisciplinary multimodal integrated care program in patients with chronic migraine and/or tension-type headache.

158 patients with chronic migraine or tensions-type headache at least five days per month for at least 6 months and current intake of triptans (migraine) or analgesic drugs (tension-type headache) are eligible. Patients undergo inpatient, outpatient and/or semi-stationary treatment including conventional headache diagnostics and therapy as well as traditional Chinese medicine, European naturopathy, and mind-body-medicine approaches. Headache frequency is defined as the primary outcome; secondary outcomes include pain (visual analog scale, Pain Perception Scale), triptans and analgesics use (headache diary), health-related quality of life (SF-36), function (Headache Disability Inventory, Patient-specific Functional Scale), depression and anxiety (Hospital Anxiety and Depression Scale), and pain self-efficacy (Pain Self-Efficacy Questionnaire). Outcomes are assessed at treatment start, treatment end and 6 months after treatment end.

DETAILED DESCRIPTION:
Chronic headache is among the most common neurological disorders with major physical, psychological, social and economic impact. The aim of this prospective observational study isto investigate the effects of an interdisciplinary multimodal integrated care program in patients with chronic migraine and/or tension-type headache.

158 patients with chronic migraine or tensions-type headache at least five days per month for at least 6 months and current intake of triptans (migraine) or analgesic drugs (tension-type headache) are eligible. Patients undergo inpatient, outpatient and/or semi-stationary treatment including conventional headache diagnostics and therapy as well as traditional Chinese medicine, European naturopathy, and mind-body-medicine approaches. Headache frequency is defined as the primary outcome; secondary outcomes include pain (visual analog scale, Pain Perception Scale), triptans and analgesics use (headache diary), health-related quality of life (SF-36), function (Headache Disability Inventory, Patient-specific Functional Scale), depression and anxiety (Hospital Anxiety and Depression Scale), and pain self-efficacy (Pain Self-Efficacy Questionnaire). Outcomes are assessed at treatment start, treatment end and 6 months after treatment end.

ELIGIBILITY:
Inclusion Criteria:

headache at least five days per month for at least 6 months current intake of a) at least 10 triptans per month or b) analgesic drugs that can themselves elicit headache

Exclusion Criteria: None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients insured with Barmer GEK or Techniker Krankenkasse, large German statutory health insurances, and diagnosed with migraine and/or tension-type headaches were eligible for integrated care. All patients, who were over 18 years old with headache at least five days per month for at least 6 months and current intake of a) at least 10 triptans per month or b) analgesic drugs that can themselves elicit headache were suited to be involved in the observational study. Patients were referred by specialists or general practitioners to the Department of Internal and Integrative Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2011-08-18 (Actual); Primary Completion 2013-07-30 (Actual); Study Completion 2014-01-30 (Actual)

PRIMARY OUTCOMES:
Headache frequency | Treatment end, an average of 5 months
  Headache days/month

SECONDARY OUTCOMES:
Headache frequency | 6 months after treatment end
  Headache days/month
Pain intensity | Treatment end, an average of 5 months
  100mm visual analog scale
Pain intensity | 6 months after treatment end
  100mm visual analog scale
Pain bothersomeness | Treatment end, an average of 5 months
  100mm visual analog scale
Pain bothersomeness | 6 months after treatment end
  100mm visual analog scale
Pain perception | Treatment end, an average of 5 months
  Pain Perception Scale
Pain perception | 6 months after treatment end
  Pain Perception Scale
Quality of life | Treatment end, an average of 5 months
  SF-12
Quality of life | 6 months after treatment end
  SF-12
Headache Disability | Treatment end, an average of 5 months
  Headache Disability Inventory (HDI)
Headache Disability | 6 months after treatment end
  Headache Disability Inventory (HDI)
Anxiety/Depression Scale | Treatment end, an average of 5 months
  Hospital Anxiety and Depression Scale (HADS)
Anxiety/Depression Scale | 6 months after treatment end
  Hospital Anxiety and Depression Scale (HADS)
Function | Treatment end, an average of 5 months
  Patient-specific Functional Scale (PSFS)
Function | 6 months after treatment end
  Patient-specific Functional Scale (PSFS)
Self-Efficacy | Treatment end, an average of 5 months
  Pain Self-Efficacy Questionnaire (FESS)
Self-Efficacy | 6 months after treatment end
  Pain Self-Efficacy Questionnaire (FESS)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No